CLINICAL TRIAL: NCT01033396
Title: A Randomized, Double Blind, Placebo Controlled, Four Way Crossover Study To Determine The Effects Of PF-03654764 +/- Allegra (Fexofenadine) On Symptoms Of Allergic Rhinitis In Subjects Exposed To Ragweed Pollen In An Environmental Exposure Unit.
Brief Title: The Effect Of PF-03654764 +/- Allegra On Symptoms Of Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B0711005
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis Environmental exposure unit
MeSH Terms: conditions — Rhinitis, Allergic | interventions — 3-fluoro-3-(3-fluoro-4-(pyrrolidin-1-ylmethyl)phenyl)-N-(2-methylpropyl)cyclobutanecarboxamide; fexofenadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-03654764 + Allegra (Experimental)
  Interventions: Drug: PF-03654764; Drug: Allegra
- PF-03654764 (Experimental)
  Interventions: Drug: PF-03654764
- Allegra-D (Active Comparator)
  Interventions: Drug: Allegra-D
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-03654764 — PF-03654764 single dose 5 mg
  Arms: PF-03654764 + Allegra
Drug: Allegra — Fexofenadine single dose 60 mg
  Arms: PF-03654764 + Allegra
Drug: PF-03654764 — PF-03654764 single dose 5 mg
  Arms: PF-03654764
Drug: Allegra-D — Fexofenadine 60 mg combined with pseudoephedrine 120 mg single dose
  Arms: Allegra-D
Drug: Placebo — Placebo single dose
  Arms: Placebo

SUMMARY:
PF-03654764 should reduce the symptoms of allergic rhinitis. In this study patients will be exposed to pollen and their symptoms observed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18-60 years allergic to ragweed pollen.
* Subjects with appropriate symptom scores following exposure to ragweed in the environmental exposure unit.

Exclusion Criteria:

* Subjects with significant diseases other than allergic rhinitis that may interfere with the safety or efficacy of PF-03654764.
* Subjects with significant symptoms of allergic rhinitis within the 2 weeks prior to screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Congestion scores | 6 hours
Other allergic rhinitis symptoms | 6 hours

SECONDARY OUTCOMES:
Pharmacokinetics | 6 hours
Blood pressure/pulse rate | 6 hours
Adverse event reporting | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Kingston, Ontario, Canada

REFERENCES:
- [Derived] North ML, Walker TJ, Steacy LM, Hobsbawn BG, Allan RJ, Hackman F, Sun X, Day AG, Ellis AK. Add-on histamine receptor-3 antagonist for allergic rhinitis: a double blind randomized crossover trial using the environmental exposure unit. Allergy Asthma Clin Immunol. 2014 Jul 3;10(1):33. doi: 10.1186/1710-1492-10-33. eCollection 2014. PMID 25024716
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0711005&StudyName=The%20Effect%20Of%20PF-03654764%20+/-%20Allegra%20On%20Symptoms%20Of%20Allergic%20Rhinitis